CLINICAL TRIAL: NCT02796534
Title: Prevalence of Obstructive Sleep Apnea Syndrome in Type 1 Diabetic Patients Treated With Insulin Pump (At1Home)
Acronym: AT1Home
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: VitalAire (Industry); ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: 38RC14.199
Record Dates: First submitted 2016-05-23; First posted 2016-06-10 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Diagnosis of sleep apnea by oxymetry

SUMMARY:
Patients with type 1 diabetes have poorer glycemic control that could lead to macrovascular or neuropathic complications; in addition to an optimal treatment, prevention of diabetes complications requires to control associated risk factors, such as hypertension or dyslipidemia. Sleep apnea syndrome is a public health problem due to its high prevalence and marked morbidity and mortality, one increasingly interesting aspect is its relationship with metabolic disorders, specifically diabetes.Obstructive sleep apnea syndrome seems to be underestimated in this population. In this context, it appears to be important to estimate the prevalence of sleep respiratory diseases in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years
* Type 1 diabetic
* Treated on insulin therapy by external pump
* Take home monitoring as part of a usual care for insulin therapy by external pump
* Voluntary to participate in research with written informed consent
* Patient affiliated to the social security or similar regime

Exclusion Criteria:

Privited person of liberty by judicial or administrative decision, person covered by legal protection (pregnant or lactating women, patients under guardianship) Article L1121-8

* In exclusion period of other studies
* Patient may, at the discretion of the investigator, not comply with the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 patients treated by Insulin Pump.
Sampling Method: Non-Probability Sample
Enrollment: 825 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea syndrome by oxymetry, confirmed by polysomnography | 2 years
  Number of patients presenting an obstructive apnea syndrome

SECONDARY OUTCOMES:
Relationship between sleep apnea syndrome severity and micro/macro vascular complications of type 1 diabetes | 2 years
  Number and type of micro and macro vascular complications will be analysed from medical history and new events will be collected at each visit and validated by endocrinologist
Relationship between sleep apnea syndrome severity and type 1 diabetes control | 2 years
  Results from regularly prescribed HbA1c analysis will be collected
Compliance of the Continuous Positive Airway Pressure (CPAP) after 3 months of use in patients with type 1 diabetes treated for severe SAS. | 2 years
  Objective compliance to the CPAP treatment is daily recorded into the device and will be provided by home care provider
Incidence of new cardiovascular events and changes in microangiopathic complications of diabetes patients depending on the presence of sleep apnea syndrome and to the adherence to CPAP treatment in case of sleep apnea syndrome treated | 2 years
  New events will be collected by asking the patients, after 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Md, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pepin JL, Bailly S, Texereau JB, Sonnet E, Picard S, Verges B, Coffin Boutreux C, Arnault Ouary G, Kessler L, Guerci B, Anton Kuchly B, Fendri Gaied S, Cuperlier A, Voinot C, Derrien C, Dubois S, Lavergne F, Borel AL, Tamisier R, Benhamou PY. Prevalence of sleep apnoea in patients with type 1 diabetes and its association with comorbidities and diabetic complications: A French nationwide prospective study. Diabetes Obes Metab. 2023 Jun;25(6):1624-1631. doi: 10.1111/dom.15015. Epub 2023 Mar 3. PMID 36792920